CLINICAL TRIAL: NCT03906474
Title: A Clinical Study to Assess the Safety of Primary, Secondary and Tertiary Blood-stage Controlled Human Plasmodium Falciparum Malaria Infection of Healthy Malaria-naïve UK Adults, and to Characterise Parasite Growth Dynamics
Brief Title: VAC063C: A Study to Assess Repeat Blood-stage P. Falciparum Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VAC063C
Record Dates: First submitted 2018-10-08; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): A third blood-stage controlled human P. falciparum malaria infection will be administered to individuals who have previously been exposed to two blood-stage challenges in the VAC063 trial. Group 1 will be challenged in parallel with Groups 2 (undergoing a second challenge) and 3 (malaria-naïve controls).
  Interventions: Biological: Blood-stage controlled human P. falciparum malaria infection
- Group 2 (Experimental): A second blood-stage controlled human P. falciparum malaria infection will be administered to individuals who have previously been exposed to one blood-stage challenge in the VAC063 trial. Group 2 will be challenged in parallel with Groups 1 (undergoing a third challenge) and 3 (malaria-naïve controls).
  Interventions: Biological: Blood-stage controlled human P. falciparum malaria infection
- Group 3 (Experimental): Malaria-naïve controls will receive a primary blood-stage controlled human P. falciparum malaria infection. Group 3 will be challenged in parallel with Groups 1 (undergoing a third challenge) and 2 (undergoing a second challenge).
  Interventions: Biological: Blood-stage controlled human P. falciparum malaria infection

INTERVENTIONS:
Biological: Blood-stage controlled human P. falciparum malaria infection — Volunteers will be challenged with malaria by administering a small amount of P. falciparum infected blood intravenously.

SUMMARY:
This is a clinical study to assess the safety of primary, secondary and tertiary blood-stage controlled human Plasmodium falciparum malaria infection of healthy malaria-naïve UK adults, as well as to evaluate any effect of prior exposure to a blood-stage controlled human malaria infection (CHMI) on the parasite multiplication rate.

As a secondary objective, the immune response to primary, secondary and tertiary P. falciparum blood-stage infection, as well as gametocytaemia, will also be assessed.

DETAILED DESCRIPTION:
Nine to seventeen healthy adult volunteers, aged between 18 and 50 years, will be recruited and receive a blood-stage controlled human malaria infection (CHMI) at the CCVTM, Oxford. Of these volunteers, three will be newly recruited, malaria-naïve volunteers, who will receive a primary CHMI.

The remaining volunteers will be invited to be involved in this study, following previous participation in the VAC063 study (ClinicalTrials.gov Identifier: NCT02927145). VAC063 was a study to assess the safety, immune responses and efficacy of the new malaria vaccine RH5.1/AS01. As part of this study, control volunteers, who did not receive a vaccine, received a blood-stage CHMI, or "challenge", in order to compare to the vaccinated volunteers. Some control (unvaccinated) participants received two challenges and some received just one challenge, therefore, in this study, participants who previously took part in VAC063 will receive either a third or second malaria challenge.

Volunteers will be challenged with malaria by administering a small amount of P. falciparum infected blood intravenously. Blood will then be taken at regular intervals to measure the parasite growth, quantify the sexual parasite forms and assess the immune response to primary, secondary or tertiary P. falciparum CHMI.

When volunteers are diagnosed with malaria, treatment with a standard antimalarial course of oral artemether-lumefantrine (Riamet) will be given over 3 days.

Volunteers who take part in this study will be involved in the trial for approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner (GP).
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and on the day prior to blood-stage CHMI, and prior to the start of antimalarial treatment.
* Provide written informed consent.
* Agreement to permanently refrain from blood donation, as per current UK Blood Transfusion and Tissue Transplantation Services guidelines.
* Reachable (24 hours a day) by mobile phone during the period between CHMI and completion of antimalarial treatment.
* Willingness to take a curative anti-malarial regimen following CHMI.
* Answer all questions on the informed consent questionnaire correctly.
* For Groups 1-2: completion of primary or secondary challenge in the VAC063 trial, curative anti-malarials and follow-up (up until at least the C+28 visit).

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator.
* Administration of immunoglobulins and/or any blood products at any time in the past.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* History of malaria chemoprophylaxis within 30 days prior to CHMI.
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* History of allergic disease or reactions likely to be exacerbated by malaria infection.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Seropositive for hepatitis B surface antigen (HBsAg) at screening.
* Seropositive for HIV virus (antibodies to HIV) at screening
* Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* History of clinical malaria (any species - NOT applicable to prior challenge in VAC063 study for Groups 1 and 2).
* Travel to a malaria endemic region during the study period or within the previous six months.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

Inability of the study team to contact the volunteer's GP to confirm medical history to allow Investigator to assess safety to participate.

* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait or any haematological condition that could affect susceptibility to malaria infection.
* Laboratory evidence of G6PD deficiency at screening.
* Laboratory evidence of haemoglobinopathy at screening.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Contraindications to the use of both Riamet and Malarone.
* Any clinical condition known to prolong the QT interval.
* Family history of congenital QT prolongation or sudden death.
* Positive family history in both 1st and 2nd degree relatives < 50 years old for cardiac disease.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Volunteer unable to be closely followed for social, geographic or psychological reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
The safety of primary, secondary and tertiary blood-stage controlled human Plasmodium falciparum malaria infection of healthy malaria-naïve UK adults, as measured by (S)AE occurrences. | 3 months
The effect of prior blood-stage CHMI on parasite multiplication rate following tertiary (Group 1) and secondary (Group 2) homologous CHMI in unvaccinated volunteers, compared to primary challenge in new malaria naïve controls (Group 3). | 3 months
  The qPCR-derived parasite multiplication rate (PMR) will be the primary endpoint for the trial, and reporting of the endpoint for Groups 1-3 will constitute the primary analysis.

SECONDARY OUTCOMES:
P. falciparum specific immunogenicity following primary, secondary and tertiary P. falciparum blood-stage infection, as assessed by antibody, B cell and T cell responses | 2 years
Gametocytaemia following primary, secondary and tertiary P. falciparum blood-stage infection. | 2 years
  Gametocytaemia will be measured by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, MBBS MA DPhil MRCP FRCPath, Principal Investigator — University of Oxford
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Salkeld J, Themistocleous Y, Barrett JR, Mitton CH, Rawlinson TA, Payne RO, Hou MM, Khozoee B, Edwards NJ, Nielsen CM, Sandoval DM, Bach FA, Nahrendorf W, Ramon RL, Baker M, Ramos-Lopez F, Folegatti PM, Quinkert D, Ellis KJ, Poulton ID, Lawrie AM, Cho JS, Nugent FL, Spence PJ, Silk SE, Draper SJ, Minassian AM. Repeat controlled human malaria infection of healthy UK adults with blood-stage Plasmodium falciparum: Safety and parasite growth dynamics. Front Immunol. 2022 Aug 22;13:984323. doi: 10.3389/fimmu.2022.984323. eCollection 2022. PMID 36072606